CLINICAL TRIAL: NCT00425282
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of RWJ-333369 as Adjunctive Therapy in Subjects With Partial Onset Seizures Followed by an Open-Label Extension Study.
Brief Title: A Study of the Efficacy and Safety of RWJ-333369 as add-on Therapy in the Treatment of Partial Onset Seizures.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR013012
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Epilepsy; Epilepsy, Focal; Seizure Disorder; Complex Partial Seizures; Epilepsy, Complex Partial
Keywords: RWJ-333369; anticonvulsants; antiepileptic drugs
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial; Seizures; Epilepsy, Complex Partial | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

INTERVENTIONS:
Drug: RWJ-333369

SUMMARY:
The purpose of this study is to demonstrate that RWJ-333369 is safe and effective as add-on treatment of partial onset seizures.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), epilepsy afflicts more than 50 million people worldwide. Despite the ongoing use of older antiepileptic drugs (AEDs) and the development of newer treatments that are better tolerated, approximately 30% of patients, particularly those with partial seizures, are not well controlled even on newer treatments, or experience significant side effects from treatment. RWJ-333369 is a drug with anticonvulsant activity that is being investigated for the treatment of epilepsy. This is a randomized (patients are assigned different treatments based on chance), double-blind study (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage ) in males and females who have partial onset seizures that have had an inadequate response to at least one AED. The study consists of 3 phases: pretreatment (a screening visit and a 56-day baseline period), double-blind treatment (12 weeks of treatment with either 200 mg per day of RWJ-333369, 400 mg per day of RWJ-333369, or placebo), and posttreatment (a posttreatment visit that occurs 7 to 14 days after the last dose of double-blind study drug). The posttreatment phase is only for patients not continuing in the open-label extension study. The open-label extension study is offered after completion of the double-blind treatment phase if the study doctor judges that the patient may benefit from continued treatment with RWJ-333369. The open-label extension study lasts until RWJ-333369 becomes available by prescription or its development is stopped by the sponsor. The efficacy of the RWJ-333369 will be based on a change in the frequency and severity of seizures. Safety assessments include adverse events (side effects) reporting, collecting blood tests and Electrocardiograms and performing physical exams, including vitals signs. The study hypothesis is that 400 mg per day of RWJ-333369 is better than placebo as add-on treatment of partial onset seizures, as measured by the percent reduction from baseline in the monthly partial onset seizure frequency. 200 mg per day RWJ-333369, 400 mg per day RWJ-333369, or placebo, given twice daily with or without food approximately 12 hours apart; study drug should be swallowed whole and not be chewed, divided, crushed, or dissolved.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, 16 year or older
* Clinical diagnosis of focal epilepsy for at least 1 year
* History of poor response to at least 1 anti-epileptic drug in the past
* Current treatment with 1 or 2 anti-epileptic drugs
* Should have at least 3 seizures per month

Exclusion Criteria:

* Generalized epilepsy
* Cannot count your seizures
* Unstable medical disease, such as a recent heart attack or uncontrolled diabetes
* Major psychiatric illness
* Recent drug or alcohol abuse
* Unable to swallow pills

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2006-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the change in seizure frequency of all simple partial motor, complex partial, or secondarily generalized seizures from the pretreatment baseline phase compared with the double-blind treatment phase.

SECONDARY OUTCOMES:
The key secondary outcome is the change in the Seizure Severity Questionnaire score.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Lu C, Zheng J, Cao Y, Bresnahan R, Martin-McGill KJ. Carisbamate add-on therapy for drug-resistant focal epilepsy. Cochrane Database Syst Rev. 2021 Dec 6;12(12):CD012121. doi: 10.1002/14651858.CD012121.pub2. PMID 34870321
- [Derived] Sperling MR, Greenspan A, Cramer JA, Kwan P, Kalviainen R, Halford JJ, Schmitt J, Yuen E, Cook T, Haas M, Novak G. Carisbamate as adjunctive treatment of partial onset seizures in adults in two randomized, placebo-controlled trials. Epilepsia. 2010 Mar;51(3):333-43. doi: 10.1111/j.1528-1167.2009.02318.x. Epub 2009 Oct 27. PMID 19863578